CLINICAL TRIAL: NCT06672783
Title: Impact of Focused Echocardiography in Management of Patients in Pediatric Intensive Care Units
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Doaa Hassan Ahmed, Resident-pediatric department-sohag hospital university, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: soh-Med-24-09-06MS
Record Dates: First submitted 2024-10-09; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Critical Patients in Pediatric Intesive Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: echocardiogrphy — Transthoracic echocardiography
  • Parameters assessed:
  * Right ventricular dimensions and function
  * Pulmonary artery pressure estimation
  * Valvular function assessment
  * Left ventricular dimensions (end-diastolic and end-systolic)o Left ventricular function (ejection fraction, fractional shortening) o

SUMMARY:
Echocardiography is currently considered a key tool for the hemodynamic assessment in Intensive Care Units (ICU), able to identify causes of hemodynamic instability and to quickly guide therapy . Some of its advantages are being a noninvasive method, risk-free, capable of being performed serially and in real time, and analyzed along with clinical data by intensivists. Several studies have demonstrated the positive effect of the use of echocardiography in the management of critically ill patients, changing their treatment in 30%-60% of cases after the test is performed . Echocardiography has been used as an adjunct in predicting patient outcomes. Relevant and easily obtain-able information about hemodynamics is required for effective therapeutic manipulation of circulation in critically ill children ,Hemodynamic monitoring of critically ill infants and children noninvasively using echocardiography has been evaluated comprehensively Echocardiography is an influential procedure that allows direct visualization of the heart, guiding patients' hemodynamic condition at the bedside. This hemodynamic estimate informs physicians to guide therapeutic approaches like volume resuscitation, initiation, discontinuation, alteration of vasopressor therapy and referral for specialist rapidly if cardiac or surgical attempt is necessary Management of critically ill pediatric patients is a demanding task that requires proper prioritization and judicious time management. Multi-system affection with overlap of symptoms often complicates the clinical picture. Hemodynamic assessment has recently taken top priority in the management of critically ill patients, Echocardiography is an integral component of the clinical service in the pediatric intensive care unit (PICU). It is considered a handy bedside imaging modality, and an accurate diagnostic tool that explores a crucial body system. Indications of bedside echocardiography in TINEC (training in intensive care and neonatal echocardiography) include assessing cardiac function, pulmonary hypertension, severe pericardial effusion, and tamponade. Consequently, it serves as a guide for interventions in critically ill pediatric patients and management .

ELIGIBILITY:
Inclusion Criteria:

* All critically ill patients admitted to pediatric intensive care units aged from 1 month Up to 18 years old.

Exclusion Criteria:

* non crtical ill patients

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Impact of focused echocardiography in management of patients in pediatric intensive care units | Through study completion , an average of one year
  functional echocardiography (ejection fraction using M mode echocardiography .
Impact of focused echocardiography in management of patients in pediatric intensive care units | Through study completion , an average of one year
  Functional echocardiography (fraction shortening by M mode echocardiography .
Impact of focused echocardiography in management of patients in pediatric intensive care units | Through study completion , an average of one year
  Assessment of pulmonary hypertension using peak tricuspid regurgitation velocity by color Doppler .
Impact of focused echocardiography in management of patients in pediatric intensive care units | Through study completion , an average of one year
  assessment of myocardial performance index.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vieillard-Baron A, Prin S, Chergui K, Dubourg O, Jardin F. Hemodynamic instability in sepsis: bedside assessment by Doppler echocardiography. Am J Respir Crit Care Med. 2003 Dec 1;168(11):1270-6. doi: 10.1164/rccm.200306-816CC. No abstract available. PMID 14644922
- [Background] Croft LB, Duvall WL, Goldman ME. A pilot study of the clinical impact of hand-carried cardiac ultrasound in the medical clinic. Echocardiography. 2006 Jul;23(6):439-46. doi: 10.1111/j.1540-8175.2006.00240.x. PMID 16839380
- [Background] Manasia AR, Nagaraj HM, Kodali RB, Croft LB, Oropello JM, Kohli-Seth R, Leibowitz AB, DelGiudice R, Hufanda JF, Benjamin E, Goldman ME. Feasibility and potential clinical utility of goal-directed transthoracic echocardiography performed by noncardiologist intensivists using a small hand-carried device (SonoHeart) in critically ill patients. J Cardiothorac Vasc Anesth. 2005 Apr;19(2):155-9. doi: 10.1053/j.jvca.2005.01.023. PMID 15868520
- [Background] Ranjit S, Aram G, Kissoon N, Ali MK, Natraj R, Shresti S, Jayakumar I, Gandhi D. Multimodal monitoring for hemodynamic categorization and management of pediatric septic shock: a pilot observational study*. Pediatr Crit Care Med. 2014 Jan;15(1):e17-26. doi: 10.1097/PCC.0b013e3182a5589c. PMID 24196006